CLINICAL TRIAL: NCT05253807
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Advanced Non-Small Cell Lung Cancer With an FGFR Alteration Who Progressed on Previous Therapy (FIGHT 210)
Brief Title: Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Relapsed or Refractory Advanced Non-Small Cell Lung Cancer With an FGFR Alteration
Acronym: FIGHT-210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-210; 2021-004934-12 (EudraCT Number)
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Advanced Non-Small Cell Lung Cancer (NSCLC); fibroblast growth factor receptor (FGFR); FGFR1-3 mutations; FGFR1-3 fusions; FGFR1-3 rearrangements; squamous NSCLC; nonsquamous NSCLC; relapsed or refractory
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Acrocephalosyndactylia; Recurrence | interventions — pemigatinib; INCB 54828-101

STUDY DESIGN:
Intervention Model Description: Participants enrolled in this study will be assigned to 1 of 2 cohorts: Cohort A (squamous NSCLC) will enroll approximately 100 participants, and Cohort B (nonsquamous NSCLC) will enroll approximately 25 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Squamous NSCLC (Experimental): Participants with squamous NSCLC with known or likely FGFR1-3 driver mutations outside the kinase domain or fusions/rearrangements will receive intermittent dosing.
  Interventions: Drug: Pemigatinib
- Cohort B: Non-squamous NSCLC (Experimental): Participants with non-squamous NSCLC with known or likely FGFR1-3 driver mutations outside the kinase domain or fusions/rearrangements will receive intermittent dosing.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — 13.5 mg tablet
  Other Names: INCB 54828

SUMMARY:
This is an open-label, single arm study to study the safety, efficacy and tolerability of Pemigatinib when used on participants with squamous or nonsquamous NSCLC with a documented FGFR1-3 mutations or fusions/rearrangement who have progressed on prior therapies and have no available standard treatment options

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic NSCLC (Stage IIIB/C or IV per the AJCC Cancer Staging Manual, 8th Edition). Both squamous and nonsquamous NSCLC are eligible.
* Radiographically measurable disease (per RECIST v1.1). Tumor lesions located in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered measurable if progression has been clearly demonstrated in the lesion.
* Documentation of known/likely actionable known or likely FGFR1-3 alterations.
* Must have objective documented progression after at least 1 prior therapy, and must have no therapy available that is likely to provide clinical benefit. Participants who are intolerant of or decline the approved therapy are eligible only if they have no therapy available that is likely to provide clinical benefit.
* ECOG performance status of 0 to 2.
* Baseline archival tumor specimen (if less than 24 months from date of screening) or willingness to undergo a pretreatment tumor biopsy to obtain the specimen. Must be a tumor block or approximately 15 unstained slides from biopsy or resection of primary tumor or metastasis.
* Willingness to avoid pregnancy or fathering a child.

Exclusion Criteria

* Prior receipt of a selective FGFR inhibitor.
* Receipt of anticancer medications or investigational drugs for any indication or reason within 28 days before the first dose of pemigatinib. Participants must have recovered (≤ Grade 1 as per CTCAE v5.0 or at pretreatment baseline) from AEs from previously administered therapies (excluding alopecia).
* Concurrent anticancer therapy (eg, chemotherapy, immunotherapy, biologic therapy, hormonal therapy, or investigational therapy).
* Candidate for potentially curative surgery.
* Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to macular/retinal degeneration, diabetic retinopathy, and retinal detachment) as confirmed by ophthalmologic examination.
* Radiation therapy administered for the treatment of cancer lesions within 2 weeks before enrollment/first dose of study drug. Participants must have recovered from all radiation related toxicities, not require corticosteroids, and not have had radiation pneumonitis. Evidence of fibrosis within a radiation field from prior radiotherapy is permitted with medical monitor approval. A 1-week washout is permitted for palliative radiation to non-CNS disease.
* Untreated brain or CNS metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain or CNS metastases). Participants who have previously treated and clinically stable brain or CNS metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT scan) during the screening period, and if they are on a stable or decreasing dose of corticosteroids for at least 1 week.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Participants with defined laboratory values at screening.
* History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues such as the skin, kidney tendon, or vessels due to injury, disease, or aging in the absence of systemic mineral imbalance).
* History of hypovitaminosis D requiring supraphysiologic doses (eg, 50,000 UI/weekly) to replenish the deficiency. Vitamin D supplements are allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Veronese, MD, Study Director — Incyte Corporation
Locations (36):
- United States (7):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Miami Cancer Institute, Miami, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - University of Kentucky Hospital, Lexington, Kentucky
  - Spoknwrd Clinical Trials Inc., Easton, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
- France (2):
  - Hï¿½PITAL NORD - CHU MARSEILLE, Marseille
  - Chu de Toulouse Hopital Larrey Centre de Reference Des Maladies Rares de La Peau Service de Dermatol, Toulouse
- Germany (4):
  - Zentralklinik Bad Berka Gmbh, Bad Berka
  - Lungenklinik Hemer, Hemer
  - Lki Lungenfachklinik Immenhausen, Immenhausen
  - University Hospital Mannheim, Mannheim
- Italy (8):
  - Irccs Centro Di Riferimento Oncologico, Aviano
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga Orbassano, Orbassano
  - Azienda Ospedaliera Di Perugia - Ospedale Santa Maria Della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena Irccs, Roma
  - Irccs Istituto Clinico Humanitas, Rozzano
- Spain (15):
  - Complejo Hospitalario Universitario A Coruna, A Coru?a
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Ico Girona Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Ico Institut Catala D Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 8 study centers in Spain, Italy, France, and the United States.
Groups:
- Cohort A: Squamous NSCLC: Participants with squamous non-small cell lung cancer (NSCLC) with known or likely fibroblast growth factor receptor 1, 2, or 3 (FGFR1-3) driver mutations outside the kinase domain or fusions/rearrangements self-administered pemigatinib 13.5 milligrams (mg) (starting dose) as a once daily (QD) oral treatment on a 21-day cycle. Participants took study drug every day on an intermittent dose regimen (2 weeks on treatment, followed by no study drug for 1 week [dose holiday]), until documented disease progression or unacceptable toxicity was reported.
- Cohort B: Nonsquamous NSCLC: Cohort B: Nonsquamous NSCLC (Experimental) Participants with nonsquamous NSCLC with known or likely FGFR1-3 driver mutations outside the kinase domain or fusions/rearrangements, including participants who had relapsed on prior targeted therapy, self-administered pemigatinib 13.5 mg (starting dose) as a QD oral treatment on a 21-day cycle. Participants took study drug every day on an intermittent dose regimen (2 weeks on treatment, followed by no study drug for 1 week [dose holiday]), until documented disease progression or unacceptable toxicity was reported.
Period: Overall Study
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Started | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5
Not completed — Death | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Cohort A
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or a partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Response was determined by an Independent Central Radiology (ICR) review. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 267 days
Population: Full Analysis Population: all enrolled participants who received at least 1 dose of pemigatinib. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort B: Nonsquamous NSCLC: Participants with nonsquamous NSCLC with known or likely FGFR1-3 driver mutations outside the kinase domain or fusions/rearrangements, including participants who had relapsed on prior targeted therapy, self-administered pemigatinib 13.5 mg (starting dose) as a QD oral treatment on a 21-day cycle. Participants took study drug every day on an intermittent dose regimen (2 weeks on treatment, followed by no study drug for 1 week [dose holiday]), until documented disease progression or unacceptable toxicity was reported.
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 3 | 0
percentage of participants | 33.3 [0.84 to 90.57] |

2. Secondary Outcome: ORR in Cohort B
Description: ORR was defined as the percentage of participants who achieved a CR or PR based on RECIST v1.1. Response was determined by an ICR review. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 80 days
Population: Full Analysis Population. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 0 | 5
percentage of participants |  | 0.0 [0.00 to 52.18]

3. Secondary Outcome: Progression-free Survival (PFS) in Cohort A
Description: PFS was defined as the time from the first dose of study treatment until progressive disease (PD) (according to RECIST v1.1 as assessed by an ICR review) or death, whichever occurred first. PD was defined as the progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 267 days
Population: Full Analysis Population. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 3 | 0
months | 8.31 [5.19 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |

4. Secondary Outcome: Duration of Response (DOR) in Cohort A
Description: DOR was defined as the time from the date of the first CR or PR until the date of the first PD (according to RECIST v1.1 as assessed by an ICR review) or death, whichever occurred first. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 182 days
Population: Full Analysis Population. Only those participants with available data were analyzed. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 1 | 0
months | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |

5. Secondary Outcome: Overall Survival (OS) in Cohort A
Description: OS was defined as the time from the first dose of study treatment to death of any cause.
Time Frame: up to 267 days
Population: Full Analysis Population. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 3 | 0
months | NA [5.19 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died. |

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib.
Time Frame: up to 302 days
Population: Safety Population: all enrolled participants who received at least 1 dose of pemigatinib
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 3 | 5
Participants | 3 | 5

7. Secondary Outcome: Number of Participants With Any Treatment-related TEAE According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib. The investigator assessed the relationship between study drug and each occurrence of each AE/serious adverse event.
Time Frame: up to 302 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC
Number analyzed (Participants) | 3 | 5
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: up to 302 days
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events that were reported for the first time or the worsening of pre-existing events after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib, have been reported for members of the Safety Population.
Groups:
- Total: Total
Arm/Group | Cohort A: Squamous NSCLC | Cohort B: Nonsquamous NSCLC | Total
All-Cause Mortality (participants affected / at risk) | 1/3 | 4/5 | 5/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/5 | 2/8
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Squamous NSCLC (N=3) | Cohort B: Nonsquamous NSCLC (N=5) | Total (N=8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Squamous NSCLC (N=3) | Cohort B: Nonsquamous NSCLC (N=5) | Total (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 1 (5)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (8) | 3 (3) | 5 (11)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (3) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 2 (2) | 4 (5)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (3)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (3)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT05253807/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT05253807/SAP_001.pdf